CLINICAL TRIAL: NCT01411735
Title: Evaluation of Enalapril Versus Placebo in Patients With Diastolic Heart Failure
Acronym: PIE-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AG018915-01 (NIH)
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2011-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Enalapril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enalapril (Active Comparator): 2.5mg titrated up to 10mg- twice daily
  Interventions: Drug: Enalapril
- placebo (Placebo Comparator): 2.5 mg titrate up to 10mg twice daily placebo comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Enalapril — 2.5mg titrated up to 10mg twice daily
  Arms: Enalapril
Drug: placebo — 2.5mg titrated up to 10mg twice daily.
  Arms: placebo

SUMMARY:
BACKGROUND: Exercise intolerance is the primary symptom in older patients with heart failure and preserved ejection fraction (HFPEF), however little is known regarding its mechanisms and therapy.

METHODS: 71 elderly stable, compensated HFPEF patients (age 70+1 years; 80% women) with controlled blood pressure were randomized into a 12 month follow-up (FU) double-blind trial of enalapril 20 mg per day (E) vs. placebo (P). Assessments included: peak exercise oxygen consumption (VO2); six-minute walk test; Minnesota Living with HF Questionnaire (MLHF); MRI; Doppler-echocardiography; and vascular ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be 60 years of age or older.

Exclusion Criteria:

1. systolic dysfunction
2. patients with evidence of significant ischemic or valvular heart disease
3. chronic pulmonary disease.

Participants who appear preliminarily eligible are invited to a formal screening visiting with an investigator cardiology physician. They also undergoing a rest and exercise electrocardiogram and echocardiogram and pulmonary function testing as well as blood hematology and chemistry tests.

Final eligibility will be based upon all information available at the conclusion of the screening visits test, including hospital and outpatient records, history, physical examination, echocardiogram and exercise test.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2003-07; Primary Completion 2004-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
exercise capacity and aortic distensibility | 9 months
  MRI and expired gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W Kitzman, MD, Principal Investigator — Professor of Medicine-Cardiology Section